CLINICAL TRIAL: NCT04577911
Title: Using the Brain to Reveal Mental Representations of Subjective Connection
Brief Title: How is Social Connection Represented in the Brain?
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAU7311; 1R01MH125406-01 (NIH)
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Loneliness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Basic Science Experiment — participants complete cognitive tasks while undergoing functional magnetic resonance imaging (fMRI)

SUMMARY:
Nearly half of the U.S. population sometimes or always experiences loneliness, which is alarming given that loneliness confers risk for negative mental and physical health outcomes. Extensive research suggests loneliness is characterized by subjective isolation: many lonely individuals maintain a number of relationships but still report feeling lonely. The goal of this proposal is to use functional magnetic resonance imaging to reveal how the brain represents our subjective connection to and isolation from other people, which will ultimately inform optimal ways to intervene to reduce loneliness.

DETAILED DESCRIPTION:
Extensive research suggests loneliness is characterized by subjective isolation: many lonely individuals maintain a number of relationships but still report feeling lonely. Thus, a neurobiological account of loneliness requires that we understand how the brain represents subjective connections to others and how loneliness alters these representations. The long-term goal of this proposal is to identify how subjective isolation is represented in the brain in order to identify novel ways to intervene on this representation to attenuate loneliness. This study proposes that the brain organizes representations of people based on subjective connection to them, and that loneliness systematically alters this organization. The Specific Aim 1 will determine whether subjective closeness organizes self and other representations in the brain. While undergoing fMRI, participants will complete tasks in which they reflect on themselves and other people. They will also report on their subjective closeness to the other people. The study will test whether the brain organizes mental representations of the self and one's own social network members based on subjective closeness. The Specific Aim 2 will determine how loneliness modulates self and other representations in the brain. The Specific, Exploratory Aim 3 will determine the cognitive consequences of altered self and other representation in loneliness. The proposal of this study is imperative for ultimately revealing neurocognitive mechanisms to intervene on to reduce loneliness.

ELIGIBILITY:
Inclusion Criteria:

* safe for MRI scanning
* not taking psychiatric medication

Exclusion Criteria:

* not safe for MRI scanning
* taking psychiatric medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be between the ages of 18 and 65
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygenated-Level Dependent (BOLD) Response | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Meyer, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided